CLINICAL TRIAL: NCT03636412
Title: Improving Frailty With a Rigorous Ambulation Intervention in Lung Transplant Patients
Acronym: iFRAIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-529
Record Dates: First submitted 2018-08-13; First posted 2018-08-17 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Transplant-Related Disorder; Frail Elderly Syndrome; Sarcopenia; Lung Graft Dysfunction; Mobility Limitation
Keywords: lung transplant; frailty
MeSH Terms: conditions — Sarcopenia; Mobility Limitation; Frailty | interventions — Walking

STUDY DESIGN:
Intervention Model Description: Patients will be recruited pre-transplant but on re-evaluation post-transplant based on mobility post-transplant will be enrolled in the ambulatory intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ambulatory Intervention (Experimental): Patients who score greater than or equal to 6 on the John's Hopkins Highest Level of Mobility (JH-HLM) scale, up to 72 hours after transfer from the ICU to the regular nursing floor will be enrolled in an ambulatory intervention. Care technicians will ambulate patients three times per day at their level of physical ability. They will also receive physical therapy standard of care.
  Interventions: Other: Ambulation
- No Ambulator (No Intervention): Patients who score less than 6 on the John's Hopkins Highest Level of Mobility (JH-HLM) scale, up to 72 hours after transfer from the ICU to the regular nursing floor will not be enrolled in the ambulatory intervention. They will receive physical therapy standard of care.

INTERVENTIONS:
Other: Ambulation — An ambulator will walk with a patient three times a day, based on physical therapy recommendations.
  Arms: Ambulatory Intervention

SUMMARY:
The objective of this study is to assess the feasibility and effectiveness of dedicated ambulator-assisted physical activity in lung transplant inpatients. The primary hypothesis is that an ambulator-assisted intervention for lung transplant patients will prove feasible and may result in improved frailty, hospital outcomes, including less need for inpatient rehabilitation and shorter length of stay in the hospital.

DETAILED DESCRIPTION:
Lung transplant is a lifesaving intervention for patients with advanced lung disease. In addition to this, patients can experience an improved quality of life and reduction in disability post transplant. Despite extensive candidate evaluation and pre-transplant scoring, waitlist mortality remains relatively high, in 2015 at 16.4 per 100 waitlist years and post-transplant 1-year mortality 16.6%.

Frailty is defined as a "generalized vulnerability to stressors" resulting from an accumulation of cognitive and physiologic deficits, which can lead to a significant decline in health following an additional stressor such, i.e. major surgery. Frailty has been associated with delayed graft function and mortality in kidney transplant recipients and waitlist mortality in liver transplant candidates. Components of frailty include weight loss, exhaustion (self-reported), weakness, slow walking speed and low physical activity, however all these components have a complex interplay.

In lung transplant, frailty was also found to be independently associated with patient-reported disability and with subsequent de-listing or death before transplant. There is conflicting evidence regarding the role of pre-transplant frailty on post-transplant outcomes in regards to overall post-operative mortality and hospital length of stay. However, prospective investigations have shown improvements in frailty following lung transplant can lead to improved disability over the first year following lung transplant.

Physical therapy interventions aimed at elderly, frail non-transplant population, were found to be successful at reducing future frailty and mobility related disability. Important components of these regimens include resistance and endurance building exercises to improve maximum oxygen consumption and muscular strength. Identifying at-risk candidates pre- and post-transplant may allow for interventions to improve outcomes. It may also assist in preventing re-admissions, since previous investigations have shown frailty was associated with 30-day hospital re-admissions in patients with after colorectal surgery.

Post-transplant, standard care should include physical activity for patients to help prevent post-operative atelectasis, increase energy, fuel appetite and reduce frailty. In lung transplant patients, exercise following transplantation has been shown to beneficial for muscular strength, six-minute walk distance and self-reported physical functioning. However the reality of care is that physical therapy availability may limit patients from ambulating more than once daily while hospitalized. An improvement in the level of activity available to patients is critical to daily their daily progress after transplant.

The investigators hypothesize that a graded protocol of ambulation which can be implemented by a dedicated patient care nursing assistant (PCNA) multiple times daily will provide significant benefit to patients without the labor and cost requirements of full-time nursing and physical therapy expertise.

The investigators believe this intervention will improve frailty in participants. These benefits will be objectively measured with evaluation of frailty during the pre- and post-transplant period, along with documentation of hospital length of stay, discharge disposition, overall mortality, 30-day readmission rate, and the number of inpatient falls.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria (pre-transplant):

1. Participant has personally signed and dated informed consent form indicating understanding of all pertinent aspects of the study.
2. Speaks fluent English
3. Active on the waiting list for a single or bilateral lung transplant
4. Able to ambulate pre-transplant (not bed/wheelchair bound) with or without assistive device

Inclusion Criteria (post-transplant)

1. Have undergone a single or bilateral lung transplant
2. Admitted to the transplant floor (J82) after discharge from the ICU
3. Complete history and physical examination on file
4. Physical therapy consult ordered (standard of care) and JH-HLM Scale of greater than or equal to 6 within 72 hours of transfer to the transplant floor

Exclusion Criteria (pre-transplant):

1. Age <18 years
2. Admitted to hospital for expedited transplant work-up
3. Admitted to hospital prior to date of transplant
4. Current invasive mechanical ventilation or placement of ECMO cannula
5. Multi-organ transplant patients (liver-lung, heart-lung)

Exclusion Criteria (post-transplant)

1. Bed rest order placed
2. Requiring invasive mechanical ventilation during the day/night

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Hospital Length of Stay | Through study completion, approximately 1 year post-transplant
  The duration of time in days for the index admission for the patient beginning immediately after lung transplant
Regular Nursing Floor Length of Stay | Through study completion, approximately 1 year post-transplant
  The duration of time in days a patient stayed on the regular nursing floor following lung transplant
30-day readmission | Up to 30 days following discharge
  The incidence of readmission to hospital within 30 days of patient discharge from hospital after index lung transplant admission

SECONDARY OUTCOMES:
Change in physical frailty phenotype | pre-transplant to 1 year following transplant
  Change in physical frailty phenotype pre and post-transplant
Change in short physical performance battery | pre-transplant to 1 year following transplant
  Change in short physical performance battery pre and post-transplant
Change in AMPAC/6-click score | pre-transplant to 1 year following transplant
  Change in AMPAC/6-click score pre and post-transplant
Change in sarcopenia | pre-transplant to 1 year following transplant
  Change in sarcopenia pre and post-transplant (m2)
Change in nutritional status; serum albumin | pre-transplant to 1 year following transplant
  Change in nutritional status; serum albumin pre and post-transplant (g/dL)
Change in nutritional status; serum protein | pre-transplant to 1 year following transplant
  Change in nutritional status; serum protein pre and post-transplant (g/dL)
Change in nutritional status; BMI | pre-transplant to 1 year following transplant
  Change in nutritional status; BMI pre and post-transplant (kg/m2)
Change in eyeball frailty assessment | pre-transplant to 1 year following transplant
  Change in eyeball frailty assessment pre and post-transplant
Presence of aspiration | pre-transplant to 1 year following transplant
  Presence of aspiration pre and post-transplant
Readmission to ICU | Through study completion, approximately 1 year post-transplant
  Readmission to ICU during index hospitalization for lung transplant
In-hospital falls | Through study completion, approximately 1 year post-transplant
  Clinical documentation of a fall during index hospital admission for lung transplant
Aspiration event | Through study completion, approximately 1 year post-transplant
  Presence of clinical aspiration event during index hospital admission for lung transplant
Graft survival | Through study completion, approximately 1 year post-transplant
  Duration of graft functioning from transplant until patient death or re-transplantation
Accelerometer step change | pre-transplant (weeks to a year to more) and immediately after transplant, up to 1 year post-transplant
  Change in steps from pre-transplant to post-transplant
Accelerometer energy expenditure | pre-transplant (weeks to a year to more) and immediately after transplant, up to 1 year post-transplant
  Change in energy expenditure from pre-transplant to post-transplant
Accelerometer time ambulating | pre-transplant (weeks to a year to more) and immediately after transplant, up to 1 year post-transplant
  Change in time ambulating from pre-transplant to post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Marie Budev, DO, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singer JP, Singer LG. Quality of life in lung transplantation. Semin Respir Crit Care Med. 2013 Jun;34(3):421-30. doi: 10.1055/s-0033-1348470. Epub 2013 Jul 2. PMID 23821515
- [Background] Valapour M, Skeans MA, Heubner BM, Smith JM, Schnitzler MA, Hertz MI, Edwards LB, Snyder JJ, Israni AK, Kasiske BL. OPTN/SRTR 2012 Annual Data Report: lung. Am J Transplant. 2014 Jan;14 Suppl 1:139-65. doi: 10.1111/ajt.12584. PMID 24373171
- [Background] Yusen RD, Edwards LB, Kucheryavaya AY, Benden C, Dipchand AI, Dobbels F, Goldfarb SB, Levvey BJ, Lund LH, Meiser B, Stehlik J; International Society for Heart and Lung Transplantation. The registry of the International Society for Heart and Lung Transplantation: thirty-first adult lung and heart-lung transplant report--2014; focus theme: retransplantation. J Heart Lung Transplant. 2014 Oct;33(10):1009-24. doi: 10.1016/j.healun.2014.08.004. Epub 2014 Aug 14. No abstract available. PMID 25242125
- [Background] Valapour M, Skeans MA, Smith JM, Edwards LB, Cherikh WS, Uccellini K, Israni AK, Snyder JJ, Kasiske BL. OPTN/SRTR 2015 Annual Data Report: Lung. Am J Transplant. 2017 Jan;17 Suppl 1:357-424. doi: 10.1111/ajt.14129. PMID 28052607
- [Background] Singer JP, Diamond JM, Gries CJ, McDonnough J, Blanc PD, Shah R, Dean MY, Hersh B, Wolters PJ, Tokman S, Arcasoy SM, Ramphal K, Greenland JR, Smith N, Heffernan P, Shah L, Shrestha P, Golden JA, Blumenthal NP, Huang D, Sonett J, Hays S, Oyster M, Katz PP, Robbins H, Brown M, Leard LE, Kukreja J, Bacchetta M, Bush E, D'Ovidio F, Rushefski M, Raza K, Christie JD, Lederer DJ. Frailty Phenotypes, Disability, and Outcomes in Adult Candidates for Lung Transplantation. Am J Respir Crit Care Med. 2015 Dec 1;192(11):1325-34. doi: 10.1164/rccm.201506-1150OC. PMID 26258797
- [Background] Garonzik-Wang JM, Govindan P, Grinnan JW, Liu M, Ali HM, Chakraborty A, Jain V, Ros RL, James NT, Kucirka LM, Hall EC, Berger JC, Montgomery RA, Desai NM, Dagher NN, Sonnenday CJ, Englesbe MJ, Makary MA, Walston JD, Segev DL. Frailty and delayed graft function in kidney transplant recipients. Arch Surg. 2012 Feb;147(2):190-3. doi: 10.1001/archsurg.2011.1229. PMID 22351919
- [Background] McAdams-DeMarco MA, Law A, King E, Orandi B, Salter M, Gupta N, Chow E, Alachkar N, Desai N, Varadhan R, Walston J, Segev DL. Frailty and mortality in kidney transplant recipients. Am J Transplant. 2015 Jan;15(1):149-54. doi: 10.1111/ajt.12992. Epub 2014 Oct 30. PMID 25359393
- [Background] Lai JC, Feng S, Terrault NA, Lizaola B, Hayssen H, Covinsky K. Frailty predicts waitlist mortality in liver transplant candidates. Am J Transplant. 2014 Aug;14(8):1870-9. doi: 10.1111/ajt.12762. Epub 2014 Jun 16. PMID 24935609
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Wilson ME, Vakil AP, Kandel P, Undavalli C, Dunlay SM, Kennedy CC. Pretransplant frailty is associated with decreased survival after lung transplantation. J Heart Lung Transplant. 2016 Feb;35(2):173-8. doi: 10.1016/j.healun.2015.10.014. Epub 2015 Oct 19. PMID 26679297
- [Background] Singer JP, Lederer DJ, Baldwin MR. Frailty in Pulmonary and Critical Care Medicine. Ann Am Thorac Soc. 2016 Aug;13(8):1394-404. doi: 10.1513/AnnalsATS.201512-833FR. PMID 27104873
- [Background] Singer JP, Peterson ER, Snyder ME, Katz PP, Golden JA, D'Ovidio F, Bacchetta M, Sonett JR, Kukreja J, Shah L, Robbins H, Van Horn K, Shah RJ, Diamond JM, Wickersham N, Sun L, Hays S, Arcasoy SM, Palmer SM, Ware LB, Christie JD, Lederer DJ. Body composition and mortality after adult lung transplantation in the United States. Am J Respir Crit Care Med. 2014 Nov 1;190(9):1012-21. doi: 10.1164/rccm.201405-0973OC. PMID 25233138
- [Background] Jones SE, Maddocks M, Kon SS, Canavan JL, Nolan CM, Clark AL, Polkey MI, Man WD. Sarcopenia in COPD: prevalence, clinical correlates and response to pulmonary rehabilitation. Thorax. 2015 Mar;70(3):213-8. doi: 10.1136/thoraxjnl-2014-206440. Epub 2015 Jan 5. PMID 25561517
- [Background] Kelm DJ, Bonnes SL, Jensen MD, Eiken PW, Hathcock MA, Kremers WK, Kennedy CC. Pre-transplant wasting (as measured by muscle index) is a novel prognostic indicator in lung transplantation. Clin Transplant. 2016 Mar;30(3):247-55. doi: 10.1111/ctr.12683. Epub 2016 Feb 11. PMID 26701203
- [Background] Cameron ID, Fairhall N, Langron C, Lockwood K, Monaghan N, Aggar C, Sherrington C, Lord SR, Kurrle SE. A multifactorial interdisciplinary intervention reduces frailty in older people: randomized trial. BMC Med. 2013 Mar 11;11:65. doi: 10.1186/1741-7015-11-65. PMID 23497404
- [Background] Liu CK, Fielding RA. Exercise as an intervention for frailty. Clin Geriatr Med. 2011 Feb;27(1):101-10. doi: 10.1016/j.cger.2010.08.001. PMID 21093726
- [Background] Robinson TN, Wu DS, Stiegmann GV, Moss M. Frailty predicts increased hospital and six-month healthcare cost following colorectal surgery in older adults. Am J Surg. 2011 Nov;202(5):511-4. doi: 10.1016/j.amjsurg.2011.06.017. Epub 2011 Sep 3. PMID 21890098
- [Background] Wickerson L. Exercise training following lung transplant is now evidence-based practice. J Physiother. 2013 Mar;59(1):58. doi: 10.1016/S1836-9553(13)70151-6. PMID 23419920
- [Background] Langer D, Burtin C, Schepers L, Ivanova A, Verleden G, Decramer M, Troosters T, Gosselink R. Exercise training after lung transplantation improves participation in daily activity: a randomized controlled trial. Am J Transplant. 2012 Jun;12(6):1584-92. doi: 10.1111/j.1600-6143.2012.04000.x. Epub 2012 Mar 5. PMID 22390625
- [Background] Inouye SK, Wagner DR, Acampora D, Horwitz RI, Cooney LM Jr, Tinetii ME. A controlled trial of a nursing-centered intervention in hospitalized elderly medical patients: the Yale Geriatric Care Program. J Am Geriatr Soc. 1993 Dec;41(12):1353-60. doi: 10.1111/j.1532-5415.1993.tb06487.x. PMID 8227919